CLINICAL TRIAL: NCT06225739
Title: Evaluation of Electronic Pregnancy Registers and Mobile Applications as a Potential Tool for Promoting Antenatal Care and Monitoring Pregnancy Outcomes
Brief Title: Evaluation of Electronic Pregnancy Registers and Mobile Applications for Monitoring Pregnancy Outcomes ( EVAPREAP )
Status: Completed | Type: Observational
Sponsor: European Vaccine Initiative (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other); Fondation pour la Recherche Scientifique, Benin (Unknown); Groupe de Recherche Action en Sante (Other); Malawi University of Science and Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: EVAPREAP-01
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related
Keywords: Pregnancy register; Mobile application; Pregnancy outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women
  Interventions: Other: Electronic pregnancy register; Other: In-depth interviews and focus group discussions
- Health care providers: In-depth interviews (IDIs) and focus group discussions (FGDs) will be used to assess the user experience and the perceptions of pregnant women and health workers on the feasibility, usability, and acceptability of open-source mobile applications for tracking pregnancy outcomes
  Interventions: Other: In-depth interviews and focus group discussions

INTERVENTIONS:
Other: Electronic pregnancy register — Electronic pregnancy register will be created based on local ANC register to monitor pregnancy outcomes across all sites. Pregnant women of all ages attending antenatal care (ANC) facility will be registered
  Groups: Pregnant women
Other: In-depth interviews and focus group discussions — In-depth interviews (IDIs) and focus group discussions (FGDs) will be used to assess the user experience and the perceptions of pregnant women and health workers on the feasibility, usability, and acceptability of open-source mobile applications for tracking pregnancy outcomes

SUMMARY:
Monitoring pregnancy outcomes during pregnancy is very important in assessing the effectiveness of interventions. This study aims to create pregnancy registers and evaluate pregnancy mobile applications as a potential tool for monitoring pregnancy outcomes in future placental malaria (PM) vaccine trials, as well as for the implementation of any other intervention in this target group.

DETAILED DESCRIPTION:
Background: Malaria during pregnancy remains a major public health problem. A consortium from Africa and Europe is further advancing the clinical development of two PM vaccine candidates (PAMVAC-cVLP and PRIMVAC). These vaccines have previously been shown to be safe, well-tolerated and able to induce a strong and functional immune response. Monitoring pregnancy outcomes during pregnancy is very important in assessing the effectiveness of interventions against PM. The increased availability of mobile phones makes them a potential tool for improving quality of care for pregnant women, accurately collecting and reporting pregnancy outcomes in identified cohorts of pregnant women. Data on the feasibility and acceptability of the mobile applications for tracking pregnancy outcomes in the areas targeted for clinical testing of candidate PM vaccines is however limited. This study will explore the creation of electronic pregnancy registers and evaluate pregnancy mobile applications as a potential tool for monitoring pregnancy outcomes in future PM vaccine trials, as well as for the implementation of other future interventions in Ghana, Burkina Faso, Benin and Malawi.

Overall aim: To evaluate the feasibility and acceptability of open-source mobile applications in tracking pregnancy outcomes among pregnant women in sub- Saharan Africa.

Methods: The study will be carried out in two phases. The first phase will involve the mapping of health application tools, and the selection of one of the tools for the registration of pregnancies at each of the participating sites. The evaluation process will involve a two-level test namely alpha and beta. Prior to the selection of the electronic tool, the team will define the data characteristics and requirements of the pregnancy register. This will be followed by a description of the process flow and the expected functionality of the pregnancy register including visualization and reporting of outcomes of interest. After this, specifications of the interface technologies, the database technologies, and the network requirements will be determined. Each site will create a pregnancy register using REDCap. The second phase will involve the assessment of the feasibility and acceptability of mobile application. At the evaluation phase, qualitative methods will be used to assess the feasibility and acceptability of using the selected mobile application for tracking pregnancy outcomes. The selected app will be tested by pregnant women. In-depth interviews (IDIs) and focus group discussions (FGDs) will be used to explore the perceptions of pregnant women and health workers on the feasibility, usability, and acceptability of open-source mobile applications for tracking pregnancy outcomes among pregnant women. Pregnant women from rural and urban parts of the study areas who will be able to use the electronic application and are willing to participate in the interviews will be purposively selected from the pregnancy register, and health workers sampled from the health facilities.

Expected outcome: The assessment of mobile applications for monitoring pregnancy outcomes and development of pregnancy registers will build the base for future PM vaccine trials and any other interventions tackling PM. If acceptability and feasibility is demonstrated, mobile applications could be linked to other tools that will provide support to front line health care workers and patients to ensure uptake and continued access to essential maternal and neonatal care services through responsive customized needs of patients in view of routine care packages.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending ANC facility in the study area
* Pregnant women whose ANC information can be accessed at the ANC facility
* Health workers providing care to pregnant women at ANC or Maternity facilities

Exclusion Criteria:

* Pregnant women attending ANC outside the study area
* Pregnant women whose ANC information cannot be accessed at the ANC facility
* Pregnant women unwilling or unable to provide informed consent

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Phase 1 study population will include pregnant women of all ages attending antenatal care (ANC) facility. Phase 2 study population will include pregnant women aged 15-49 years attending ANC facility and health workers who provide healthcare services to pregnant women at ANC clinics or Maternity ward
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of mobile application for registration of pregnant women and tracking pregnancy outcomes | 9 months
  Assess whether an open-source mobile applications is easy and convenient to use accounting for advantages and disadvantages to guide integrating the App into routine workflow via qualitative methods: In-depth interviews (IDIs) and focus group discussions (FGDs)
Usability of mobile application for registration of pregnant women and tracking pregnancy outcomes | 9 months
  Assess whether open-source mobile applications could be used by pregnant women and health workers to adequately record, track, and summarize data, including whether it functioned in a way that enhanced productivity or led to unproductive tasks due to errors. The assessment will be done using qualitative methods: In-depth interviews (IDIs) and focus group discussions (FGDs)
Acceptability of mobile application for registration of pregnant women and tracking pregnancy outcomes | 9 months
  Acceptability will be defined as pregnant women and health workers and other stakeholders found the Client Data App acceptability, including its interface and navigation features. The assessment will be done using qualitative methods: In-depth interviews (IDIs) and focus group discussions (FGDs)

CONTACTS AND LOCATIONS:
Overall Officials: Kwaku Poku Asante, MD, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana
Locations (4):
- Fondation pour la Recherche Scientifique (FORS), Cotonou, Benin
- Groupe de Recherche Action en Santé (GRAS), Ouagadougou, Burkina Faso
- Kintampo Health Research Centre (KHRC), Kintampo, Ghana
- Malawi University of Science and Technology (MUST), Mikolongwe, Malawi

REFERENCES:
- See also: Related Info — http://www.advance-vac4pm.eu/